Symptoms Burden in Lung Cancer Patients Undergoing Definitive Chemoradiotherapy: Insights

from Electronic Patient-Reported Outcomes

Version: V1.0

Date: May 24, 2024

Principal Investigator: Dr. Qian Chu

Institution: Tongji Hospital, Tongji Medical College, Huazhong University of Science and

Technology

**Background:** 

Lung cancer remains the leading cause of cancer-related morbidity and mortality in both

men and women in China, accounting for 22.0% of new cases and 28.5% of cancer-related deaths

in 2022<sup>[1]</sup>. For patients with locally advanced non-small cell lung cancer (NSCLC) and limited-

stage small cell lung cancer (SCLC), definitive concurrent chemoradiotherapy (CRT) remains the

standard of care. Despite offering substantial local control, radiotherapy (RT) can cause adverse

events such as radiation pneumonitis, esophagitis, and dermatitis [2-4]. Radiation pneumonitis

occurs in 10-30% of patients, typically 4-12 weeks post-RT, while acute radiation esophagitis

often emerges within 2-3 weeks of treatment, significantly impairing patient quality of life.

In the era of extended survival and holistic health care, monitoring patient-reported

symptoms during CRT is crucial. Traditional clinical assessments often fail to detect moderate-to-

severe symptoms, particularly post-discharge. Therefore, a patient-centered, continuous symptom

monitoring strategy is urgently needed.

Patient-reported outcomes (PROs) are direct reports from patients about their health status

without interpretation by clinicians. These encompass symptoms, functional status, quality of life,

treatment perceptions, and adherence<sup>[5]</sup>. Electronic PROs (ePROs), which leverage smartphones

or computers, offer real-time, accurate, and scalable solutions for symptom monitoring.

In the West, ePROs are integrated into clinical trials, drug evaluations, and healthcare

quality assessments. Studies show that ePROs enhance symptom detection, improve adherence,

and prolong survival<sup>[6-9]</sup>. For example, Dr. Jennifer R. at Memorial Sloan Kettering Cancer

Center analyzed ePROs from over 12,000 surgical cancer patients, establishing postoperative

symptom trajectories. Similarly, ePRO data in metastatic HR+/HER2- breast cancer patients on oral therapy showed a reduced risk of serious adverse events<sup>[10-12]</sup>.

In China, research on ePROs is emerging. Professor Qiuling Shi's multicenter RCT implemented ePRO-based symptom monitoring in perioperative lung cancer patients, resulting in reduced complications and improved satisfaction<sup>[13]</sup>. However, no studies have yet focused on lung cancer patients receiving definitive CRT.

This study aims to evaluate symptom burden and clusters during and after CRT in lung cancer patients using validated ePRO instruments.

### **Objectives:**

To longitudinally assess symptom burden and symptom clusters among lung cancer patients undergoing definitive CRT using ePROs and to compare patterns across clinical subgroups.

### Significance:

Inform precise symptom management during and post-CRT.

Establish a PRO-driven framework for supportive care in lung cancer.

### **Study Design:**

This is a prospective observational cohort study conducted from June 2024 to December 2025 in the Department of Thoracic Oncology, Tongji Hospital. Eligible participants will be recruited prior to CRT initiation and enrolled after informed consent.

### **Primary Outcomes:**

Longitudinal trajectory of symptom burden over time based on M. D. Anderson Symptom Inventory-Lung Cancer (M. D. Anderson Symptom Inventory-Lung Cancer: Scale range 0–10, with higher scores indicating worse symptom burden)

# **Secondary Outcomes:**

- 1. Questionnaire response rate
- 2. Trajectory of symptom interference over time based on M. D. Anderson Symptom Inventory-Lung Cancer (M. D. Anderson Symptom Inventory-Lung Cancer: scale range 0–10, with higher scores indicating worse interference)

- 3. Change of Quality of life over time (Quality of life will be assessed using the EuroQoL-5 Dimension Health Outcome Survey (EQ-5D) Questionnaire, Higher scores on the EQ-5D reflect better quality of life)
- 4. Associations between symptom severity and progression-free survival (PFS).
- 5. Identification of PRO-related risk factors; development of predictive models.

# **Eligibility Criteria:**

#### **Inclusion Criteria**:

- Pathologically confirmed unresectable stage III NSCLC or limited-stage SCLC
- Age  $\geq$  18 years
- Receiving definitive concurrent chemoradiotherapy (CRT)
- Able and willing to complete electronic questionnaires
- Provided written informed consent

### **Exclusion Criteria:**

- Severe comorbidities (heart, liver, kidney)
- Psychiatric illness or cognitive impairment
- · Prior chest or mediastinal radiotherapy

# Sample Size:

Using the rule-of-thumb for factor analysis (5-10 participants per variable), with 16 symptom items, the minimum sample size is estimated at 80 patients.

# **Study Procedures:**

Participants will complete ePROs at baseline (1-2 days before CRT), weekly during CRT, and weekly for 12 weeks post-CRT.

# **Data Sources:**

EMR: Demographics, tumor characteristics, comorbidities, treatment details, labs, and costs Clinical research data platform: Survival tracking

ECOG, CTCAE v5.0: Clinical evaluations

PRO Tools:

MDASI-LC: 22 items (13 core symptoms, 3 lung-specific, 6 interference)

EQ-5D: 5 domains and visual analog scale

### **Data Collection Platform:**

WeChat mini-program with automated reminders. Trained thoracic oncology clinicians will support data entry and follow-up.

### **Risk and Ethical Considerations:**

As a non-interventional study, risks are minimal. No identifiable personal data will be collected. Study adheres to the Declaration of Helsinki.

# **Statistical Analysis:**

Mixed-effects models to analyze symptom trajectories

Descriptive statistics for symptom frequency/severity

Cox models for associations with PFS and OS

PCA, EFA, and hierarchical clustering to identify symptom clusters

Multivariate regression and nomogram development for prediction modeling

### References

- [1] Zheng RS, Chen R, Han BF, et al. [Cancer incidence and mortality in China, 2022]. Zhonghua Zhong Liu Za Zhi. 2024. 46(3): 221-231.
- [2] Hanania AN, Mainwaring W, Ghebre YT, Hanania NA, Ludwig M. Radiation-Induced Lung Injury: Assessment and Management. Chest. 2019. 156(1): 150-162.
- [3] Behroozian T, Bonomo P, Patel P, et al. Multinational Association of Supportive Care in Cancer (MASCC) clinical practice guidelines for the prevention and management of acute radiation dermatitis: international Delphi consensus-based recommendations. Lancet Oncol. 2023. 24(4): e172-e185.
- [4] Alam SR, Zhang P, Zhang SY, et al. Early Prediction of Acute Esophagitis for Adaptive Radiation Therapy. Int J Radiat Oncol Biol Phys. 2021. 110(3): 883-892.

- [5] Bennett AV, Jensen RE, Basch E. Electronic patient-reported outcome systems in oncology clinical practice. CA Cancer J Clin. 2012. 62(5): 337-47.
- [6] Hollen PJ, Gralla RJ, Liepa AM, Symanowski JT, Rusthoven JJ. Adapting the Lung Cancer Symptom Scale (LCSS) to mesothelioma: using the LCSS-Meso conceptual model for validation. Cancer. 2004. 101(3): 587-95.
- [7] Pompili C, Koller M, Velikova G, et al. EORTC QLQ-C30 summary score reliably detects changes in QoL three months after anatomic lung resection for Non-Small Cell Lung Cancer (NSCLC). Lung Cancer. 2018. 123: 149-154.
- [8] Temel JS, Greer JA, Muzikansky A, et al. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010. 363(8): 733-42.
- [9] Mendoza TR, Wang XS, Lu C, et al. Measuring the symptom burden of lung cancer: the validity and utility of the lung cancer module of the M. D. Anderson Symptom Inventory. Oncologist. 2011. 16(2): 217-27.
- [10] Cracchiolo JR, Tin AL, Assel M, et al. Electronic Patient-Reported Symptoms After Ambulatory Cancer Surgery. JAMA Surg. 2024.
- [11] Kalinsky K, Accordino MK, Chiuzan C, et al. Randomized Phase II Trial of Endocrine Therapy With or Without Ribociclib After Progression on Cyclin-Dependent Kinase 4/6 Inhibition in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer: MAINTAIN Trial. J Clin Oncol. 2023. 41(24): 4004-4013.
- [12] Li JJ, Li JR, Wu JM, et al. Change in symptom clusters perioperatively in patients with lung cancer. Eur J Oncol Nurs. 2021. 55: 102046.
- [13] Dai W, Feng W, Zhang Y, et al. Patient-Reported Outcome-Based Symptom Management Versus Usual Care After Lung Cancer Surgery: A Multicenter Randomized Controlled Trial. J Clin Oncol. 2022. 40(9): 988-996